CLINICAL TRIAL: NCT01901250
Title: Xylitol for Caries Prevention in Inner-City Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Principal Investigator, Suchitra Nelson, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11-06-18; R40MC07838 (Other Grant/Funding Number: HRSA/MCHB)
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Dental Caries
Keywords: Dental Caries; Xylitol; Prevention
MeSH Terms: conditions — Dental Caries | interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xylitol GB (Experimental): Xylitol gummy bears 7.8g/day throughout the 9 month kindergarten year, oral health education, fluoride varnish, and dental sealant
  Interventions: Dietary Supplement: Xylitol gummy bears; Behavioral: Oral health education; Device: Fluoride varnish; Device: Dental sealant
- Fiber GB (Placebo Comparator): Sugar free fiber gummy bears 20g/day throughout the 9 month kindergarten year, oral health education, fluoride varnish, and dental sealant
  Interventions: Dietary Supplement: Sugar free fiber gummy bears; Behavioral: Oral health education; Device: Fluoride varnish; Device: Dental sealant

INTERVENTIONS:
Dietary Supplement: Xylitol gummy bears — The children receive xylitol gummy bears 3 times/day within the supervised school environment.
  Arms: Xylitol GB
Dietary Supplement: Sugar free fiber gummy bears — The children receive sugar free fiber gummy bears 3 times/day within the supervised school environment.
  Arms: Fiber GB
Behavioral: Oral health education — Oral health education, toothbrush, and fluoride toothpaste
Device: Fluoride varnish — The study dentists apply the varnish on all children twice a year during the study period. The varnish is 5% sodium fluoride and contains 2.26% by weight fluoride ion in a colophony base.
  Other Names: Cavity Shield
Device: Dental sealant — The study dentists apply the sealant on the children in the second grade when the permanent first molars are fully erupted.
  Other Names: UltraSeal XT plus

SUMMARY:
The purposes of this study is to determine whether xylitol use in kindergarten school children in addition to oral health education, provision of tooth brush and fluoride paste, fluoride varnish and sealant treatment will reduce decay in the first permanent molars and other permanent teeth.

DETAILED DESCRIPTION:
This is a two group, 30 month randomized controlled clinical trial to assess, in conjunction with other primary preventive modalities, the use of xylitol gummy bears as snack food during school hours to reduce dental caries among children attending Kindergarten at the time of recruitment.

Classrooms in five elementary schools were randomized to receive xylitol gummy bears or the control sugar-free (fiber) gummy bears. All gummy bears were formulated to be similar in size, consistency, color, and sweetness. They were in six bright colors attractive to children, and in strawberry and cherry flavors which are popular among children. Children were encouraged to chew the gummy bears slowly to maximize the xylitol exposure time in the mouth. The children received xylitol or placebo gummy bears throughout the 9 month kindergarten year, 3 times/day within the supervised school environment.

In addition to gummy bears, all participating children received oral health education, tooth brushing and fluoridated toothpaste, topical fluoride varnish treatment, and dental sealants when the first permanent molars have completely erupted. This design allows for the comparison between the current best recommended public heath practices and the addition of the new strategy, xylitol gummy bear snacks. Children were enrolled in kindergarten and followed until the middle of 2nd grade.

ELIGIBILITY:
Inclusion Criteria:

* attending kindergarten in one of the participating schools
* must have parental permission

Exclusion Criteria:

* children with severe stomach illness (ex. Crohn's disease, ulcerative colitis, Celiac disease, irritable bowel syndrome, etc.)
* children with strict dietary restriction (ex. Diabetes)

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 562 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Nelson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Background] Nelson S, Eggertsson H, Powell B, Mandelaris J, Ntragatakis M, Richardson T, Ferretti G. Dental examiners consistency in applying the ICDAS criteria for a caries prevention community trial. Community Dent Health. 2011 Sep;28(3):238-42. PMID 21916361
- [Background] Nelson S, Milgrom P. Minority participation in a school-based randomized clinical trial of tooth decay prevention in the United States. Contemp Clin Trials. 2012 Jan;33(1):60-6. doi: 10.1016/j.cct.2011.09.012. Epub 2011 Oct 1. PMID 21986390
- [Background] Nelson S, Mandelaris J, Ferretti G, Heima M, Spiekerman C, Milgrom P. School screening and parental reminders in increasing dental care for children in need: a retrospective cohort study. J Public Health Dent. 2012 Winter;72(1):45-52. doi: 10.1111/j.1752-7325.2011.00282.x. Epub 2011 Oct 10. PMID 22316214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three cohorts of kindergarten children were recruited from 5 elementary schools between 2007 and 2009. A total of 32 classrooms were randomized to xylitol (16 classrooms) and placebo (16 classrooms).
Pre-assignment Details: Out of 562 children recruited, a total of 37 children did not have the baseline dental examination (13 children were transferred out of school district and 24 children were absent from the baseline dental examination).
Period: Overall Study
Arm/Group | Xylitol GB | Fiber GB
Started | 260 | 265
End of Kidergarten | 215 | 212
Start of 1st Grade | 173 | 176
End of 1st Grade | 143 | 151
Completed | 122 | 139
Not Completed | 138 | 126

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xylitol GB | Fiber GB | Total
Number analyzed (Participants) | 260 | 265 | 525
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 260 | 265 | 525
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 137 | 280
  Male | 117 | 128 | 245
Race/Ethnicity, Customized [Number; unit: participants]
  Black Non-Hispanic | 227 | 234 | 461
  White Non-Hispanic | 4 | 3 | 7
  Hispanic | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Unknown or Not reported | 27 | 26 | 53
Overall Caries Burden at Baseline [Number; unit: participants]
  None (0 dmfs/DMFS) | 112 | 138 | 250
  Moderate (1-5 dmfs/DMFS) | 68 | 66 | 134
  Severe (6 or more dmfs/DMFS) | 80 | 61 | 141

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Decayed or Filled Permanent Teeth (DFT) From Baseline (Beginning of Kindergarten) to the Middle of 2nd Grade
Description: The primary outcome measure was change in the number of decayed or filled permanent teeth (DFT). Caries was assessed in accordance to the International Caries Detection and Assessment System (ICDAS). The ICDAS criteria record both the severity and activity of the lesion on occlusal surfaces, in pit and fissure sites on the buccal and lingual surfaces, and on other smooth surfaces.
  For the purposes of this study, an ICDAS severity score of 3 to 6 and the presence of fillings constituted the "D" and "F" portions of DFT, respectively.
Time Frame: baseline and middle of 2nd grade
Measure: Mean (Standard Deviation); unit: Number of surfaces
Arm/Group | Xylitol GB | Fiber GB
Number analyzed (Participants) | 122 | 139
Number of surfaces | 0.38 (0.88) | 0.48 (1.39)
Statistical Analysis 1: Comparison: Xylitol GB vs Fiber GB; Test type: Superiority or Other; p = 0.25, Permutation test; Adjusted for child's gender, caries burden at study entry, surface-years at risk, and study cohort

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Xylitol GB | Fiber GB
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/265
Other Adverse Events (participants affected / at risk) | 0/260 | 0/265

LIMITATIONS AND CAVEATS:
Nearly half the children moved out of the school district by the time of the exit examination, which made the power of the analysis insufficient to detect the difference between two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes